CLINICAL TRIAL: NCT03801954
Title: Implementation of Nutrition Education Videos for Patients Undergoing Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00142651
Record Dates: First submitted 2018-08-02; First posted 2019-01-14 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Bladder Cancer
Keywords: Nutrition; Diet; Radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RC Patients: Patients at the University of Kansas Medical Center who have not yet had their radical cystectomy, after their radical cystectomy, or between the completion of chemotherapy and the radical cystectomy.
  Interventions: Behavioral: Educational Videos

INTERVENTIONS:
Behavioral: Educational Videos — 15 videos that are about 3 minutes long each and cover nutritional advice for patients with bladder cancer undergoing RC and/or chemotherapy.

SUMMARY:
By doing this study the investigators hope to learn if educational videos focusing on nutrition for bladder cancer patients are a good and effective way to help people improve their nutrition and recovery after radical cystectomy (RC).

DETAILED DESCRIPTION:
Bladder Cancer is the fifth most common cancer in the USA. The primary treatment for invasive bladder cancer is chemotherapy followed by RC. Patients undergoing this surgery are at risk for complications. Being malnourished can increase the risk of mortality by three times. The patients also suffer from taste alterations after chemotherapy and gastrointestinal disturbances such as diarrhea and constipation. These can lead to poor nutritional intake and malabsorption of nutrients.

This study is being done to develop an educational video series for patients undergoing RC and assess their impact. The videos are created to address the nutritional needs of these patients and improve their outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bladder cancer and scheduled to undergo a radical cystectomy or has undergone a radical cystectomy OR be the caregiver of a patient diagnosed with bladder cancer who is scheduled to undergo a radical cystectomy or has undergone a radical cystectomy

Exclusion Criteria:

* 1. Patients who are under 18 years old are not allowed to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the University of Kansas Urology clinic for bladder cancer will be screened for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate content of three educational video series | Week 2
  Evaluate the content of three video series focusing on practical solutions to nutritional problems common to patients undergoing a radical cystectomy through iterative process using Center for Disease Control's Clear Communication Index. The Center for Disease Control's Clear Communication Index uses 4 questions and 20 scored items to asses how materials enhance and aid people's understanding of information in seven areas - main message and call to action, language, information design, state of the science, behavioral recommendations, numbers, and risk. The range of scores is 0 to 100 with a score of 90 or higher considered a passing score.
Patient Feedback Regarding Videos | Week 2
  After viewing the videos semi-structure interviews of participants will be conducted to obtain feedback regarding the videos content and design.
Patient Attention During Videos | Week 2
  Eye tracking of participants will be used to assess attention of participants during the videos in order to best understand how participants are viewing the videos and responding to them.
Test feedback instrument with patients | Week 2
  Use a pretest developed instrument measuring nutrition knowledge to test participants knowledge before and after watching the videos
Assess implantation of video series | Week 2
  Online survey of viewers will be used to gain feedback on how the videos were received by those who watched them

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Lee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States